CLINICAL TRIAL: NCT00211523
Title: Phase II, Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Safety and Efficacy of MBI 226 2.5% and 5.0% Acne Solutions Applied Topically for 6 Weeks to Subjects With Acne Vulgaris
Brief Title: Safety and Efficacy of MBI 226 2.5% and 5.0% Topical Acne Solutions in the Treatment of Acne
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioWest Therapeutics Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A99004
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2005-09-21 (Estimated); Status verified 2005-09

CONDITIONS: Acne Vulgaris; Acne; Propionibacterium Acnes
Keywords: acne; acne vulgaris; MBI 226; Propionibacterium acnes; lesion counts; lesions; inflammatory; non-inflammatory; topical
MeSH Terms: conditions — Acne Vulgaris

INTERVENTIONS:
Drug: MBI 226 Acne Solutions

SUMMARY:
This study investigates the safety and efficacy of MBI 226 2.5% and 5.0% Acne Solutions, applied topically for six weeks, in the treatment of acne.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ages 13 and up, exhibiting high levels of facial P. acnes
* Presence of inflammatory and non-inflammatory lesions

Exclusion Criteria:

* Acne conglobata, acne fulminans, or secondary acne (chlorine, drug-induced acne, etc.)
* Active facial cysts

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 75
Dates: Start 2000-10; Study Completion 2001-09

PRIMARY OUTCOMES:
- percent change in inflammatory, non-inflammatory, and total acne lesion counts over entire study and dichotomized Global Severity Assessment

SECONDARY OUTCOMES:
- percent change in lesion counts after ~2 and ~4 weeks
- Global Severity Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Jim Pankovich, Study Director — BioWest Therapeutics Inc